CLINICAL TRIAL: NCT01406587
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel Group Evaluation of the Efficacy and Safety of 50 mg, 100 mg and 200 mg PP4001 Twice Daily for the Treatment of Burning During Urination, Pain, and Urination Frequency Associated With Uncomplicated Urinary Tract Infection
Brief Title: Safety and Efficacy of PP4001 for the Treatment of Symptoms Associated With Uncomplicated Urinary Tract Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pinnacle Pharmaceuticals, Inc. (Industry)
Responsible Party: Suma Krishnan, MS, MBA, Pinnacle Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PP4001.301
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Urinary Tract Infection
Keywords: Burning; Dysuria; Frequency; Pain; Uncomplicated Urinary Tract Infection; Uncomplicated UTI; Urinary Tract Infection; UTI; Burning during urination associated with uncomplicated urinary tract infection; Urination frequency associated with uncomplicated urinary tract infection; Pain associated with uncomplicated urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections; Paresthesia; Dysuria; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PP4001 50 mg (Experimental)
  Interventions: Drug: PP4001
- PP4001 100 mg (Experimental)
  Interventions: Drug: PP4001
- PP4001 200 mg (Experimental)
  Interventions: Drug: PP4001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PP4001 — 50 mg, 1 dose every 12 hours x 4 doses
  Arms: PP4001 50 mg
Drug: PP4001 — 100 mg, 1 dose every 12 hours x 4 doses
  Arms: PP4001 100 mg
Drug: PP4001 — 200 mg, 1 dose every 12 hours x 4 doses
  Arms: PP4001 200 mg
Drug: Placebo — Placebo, 1 dose every 12 hours x 4 doses
  Arms: Placebo

SUMMARY:
PP4001 is a medication not yet approved by the US FDA. This is a phase 2, multi-center, randomized, double-blind study of 3 doses of PP4001 versus placebo in the treatment of symptoms associated with uncomplicated urinary tract infection. After the screening, patients are randomized to receive one of three doses of PP4001 or placebo. Patients are screened and randomized on the same day, and take 4 doses of study drug, one dose every 12 hours. Data about uncomplicated urinary tract infection symptoms are collected from the subjects on electronic handheld devices throughout the 48-hour study period. The primary endpoint is burning during urination.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be ≥ 18 and ≤ 75 years of age at the time of consent.
* Females not of childbearing potential (FNCBP) are eligible for randomization. FNCBP are defined as postmenopausal women with their last menstrual cycle (without exogenous hormone therapy) completed more than 12 consecutive months before screening or women who are surgically sterilized (hysterectomy, oophorectomy, or tubal ligation). Females of childbearing potential also are eligible for randomization provided they are not pregnant or nursing and employ appropriate methods of contraceptives for the duration of the trial. Medically acceptable forms of contraception include abstinence, oral contraceptives, intra-uterine devices, injectable hormonals, intra-vaginal rings, or double-barrier methods (condom plus spermicide), for at least 1 month prior to treatment. Subjects in a monogamous, long term relationship with a partner who has had a vasectomy at least 3 months prior to screening are also study eligible.
* Diagnosis of uncomplicated UTI as defined by having both of the following:
* Presence of supporting symptoms including new onset (within 1 week) of urination frequency, painful urination, and/or urgency.
* Positive dipstick test for leukocyte esterase.
* Demonstration of moderate to severe burning during urination as measured by a score of at least six (6) on the 11-point rating scale for Burning During Urination during screening.
* A negative urine pregnancy test for women of childbearing potential.
* If subject has a chronic, clinically stable disease that requires medication, medication to treat that disease must be stable for at least 30 days prior to screening.
* Ability to perform study procedures, including the completion of electronic diary assessments, and supply the necessary information to the study personnel as required by the protocol.
* A signed informed consent form in which the subject agrees to participate after the study has been fully explained.

Exclusion Criteria:

* Clinically significant medical history or a clinically significant abnormal finding on the physical exam, vital signs or ECG at screening, including serious acute illness (e.g. pneumonia), gastrointestinal illness that would interfere with study drug absorption, or an untreated or unstable medical illness that would likely interfere with the study assessments.
* At risk in terms of the precautions, warnings, and contraindications in the package insert for phenazopyridine hydrochloride including:
* Known hypersensitivity to phenazopyridine hydrochloride (Defined by a history of allergic or adverse response to the drug).
* Renal failure or insufficiency (Defined as having a history of abnormal renal function or as having a known renal disease).
* History of hepatic disease or failure (Defined as having known liver disease or having elevated LFTs (> 2 times the ULN) on previous laboratory testing. Patients who would not otherwise have such testing are not required to undergo special study labs).
* Known G-6-PD (glucose-6-phosphate dehydrogenase) deficiency.
* Prior use of a phenazopyridine product within 6 months of the first dose of study drug and throughout the study.
* Use of any prescription analgesic medication (e.g. opioids, prescription nonsteroidal anti-inflammatory drugs (NSAID), etc.) for urinary tract pain or other pain (headache, back pain, joint pain, dental pain, sore muscles, etc) within one and a half (1.5) dosing intervals for that medication before the firs dose of study drug, and throughout the study.
* Use of any systemic antibiotic within seven (7) days of study participation.
* Subjects with complaint of abnormal vaginal discharge.
* Current diagnosis or suspicion of complicated UTI or systemic infection based on one or more of the following:
* Known presence of an anatomic or functional abnormality.
* Presence of a urinary catheter.
* Infection of the urinary tract requiring an intravenous pyelogram (IVP), ultrasound or cystoscopy.
* Clinical signs of systemic infection such as fever (oral or tympanic temperature >38 degrees Celsius), costovertebral pain or tenderness, rigors, nausea or vomiting.
* Subjects unable to comprehend the language of the informed consent and the self evaluation scales.
* Subjects who, in the opinion of the investigator, are not appropriate for, or are unable, or unwilling to undergo antibiotic treatment for uncomplicated urinary tract infection.
* Subjects with complaint of abnormal vaginal bleeding defined as different from the patient's usual menstrual period flow and timing.
* Subjects with known allergy to multivitamin or any component of the multivitamin.
* Currently participating in a clinical trial or has received an experimental drug or used an experimental device in the last 30 days prior to admission into this study.
* Subjects who, in the opinion of the investigator, are unsuitable for enrollment, unlikely to complete the course of study medication treatment, or unlikely to attend the End of Study visit.
* Subjects who are unable or unwilling to comply with the use of an electronic subject diary.
* Employees of the investigator or the institution who have direct involvement in the trial or other trials under the direction of the investigator or their associates.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of PP4001 for the relief of burning during urination as measured by the subject's self-reported score at the time of urination in women with uUTI in comparison to placebo. | Assessed at each urination from the time of randomization to 48 hours post first dose.

SECONDARY OUTCOMES:
Change from baseline in the physical exam evaluation at the End of Study visit | The End of Study Visit is 48 - 100 hours post first dose. SAEs will be followed up to 30 days beyond the End of Study Visit.
  Body systems evaluated will include:
  * General appearance
  * Skin
  * HEENT (Head, Ears, Eyes, Nose, Throat)
  * Spine/Neck/Thyroid
  * Respiratory
  * Cardiovascular
  * Abdomen
  * Nervous System
  * Musculoskeletal
To assess the efficacy of PP4001 for the relief of pain as measured by the subject's self-reported score at the time of urination. | Assessed at each urination from the time of randomization through 48 hours post first dose.
To assess the efficacy of PP4001 for reduction in urination frequency as measured by the subject's self-reported void diary. | Assessed at each urination from the time of randomization through 48 hours post first dose.
To evaluate the duration of therapeutic response to PP4001 50 mg, 100 mg and 200 mg. | Efficacy measures assessed in 2-hour windows after each dose.
To assess global assessment of uUTI symptom severity and change over time as measured by the subject-reported global assessment diaries. | Assessed at each urination from the time of randomization through 48 hours post first dose.
Change from baseline in vital signs at the End of Study visit | The End of Study Visit is 48 - 100 hours post first dose. SAEs will be followed up to 30 days after the End of Study Visit.
  Vital sign measures will include systolic and diastolic blood pressure, pulse, respiratory rate, and temperature.
Change from baseline in ECG at the End of Study visit | The End of Study Visit is 48 - 100 hours post first dose. SAEs will be followed up to 30 days beyond the End of Study Visit.
  ECG parameters to be reported in this study include heart rate, and interval parameters of RR, PR, QRS, QT, and QTc.
Change from baseline in laboratory evaluations at the End of Study visit | The End of Study Visit is 48 - 100 hours post first dose. SAEs will be followed up to 30 days beyond the End of Study Visit.
  The following laboratory assessments will be performed: venous blood and urine samples for clinical laboratory testing, including hematology, serum chemistry, urinalysis, and urine culture.
Frequency, severity and relationship to study medication of treatment emergent adverse events | From first dose through the End of Study Visit (48 - 100 hours post first dose)
  Frequency of treatment emergent AEs will be calculated for each body system, by preferred term, by treatment and by period for the number of subjects reporting the event for the safety population. The severity of the AEs and the relationship to study medication will be summarized for each body system and preferred term. Withdrawals due to AEs will be summarized for each body system and preferred term.

CONTACTS AND LOCATIONS:
Overall Officials: Suma Krishnan, Study Director — Pinnacle Pharmaceuticals
Locations (25):
- United States (25):
  - Drug Research and Analysis Corp., Montgomery, Alabama
  - Mesa Family Medical Center/Clincal Research Advantage, Mesa, Arizona
  - Desert Clinical Research/Clinical Research Advantage, Mesa, Arizona
  - Central Phoenix Medical Clinic/Clinical Research Advantage, Phoenix, Arizona
  - Northern California Research, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Women's Health Care Research, San Diego, California
  - Tampa Bay Medical Research, Clearwater, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Urology Center of Central Florida/Triquest Clinical Research Inc., Saint Cloud, Florida
  - Soapstone Center for Clinical Research, Decatur, Georgia
  - Hutzel Women's Health Research, Detroit, Michigan
  - Bellevue Family Practice/Clinical Research Advantage, Bellevue, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - AccuMed Research Associates, Garden City, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Hawthorne Medical Research, Inc., Winston-Salem, North Carolina
  - Hometown Urgent Care and Research, Groveport, Ohio
  - Hometown Urgent Care and Research, Springfield, Ohio
  - Ellipsis Research Group, LLC, Columbia, South Carolina
  - Palmetto Clinical Research, LLC, Greenville, South Carolina
  - InvestiClin Research, Brentwood, Tennessee
  - Advanced Research Associates, Corpus Christi, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Clinical Trials of Texas, San Antonio, Texas